CLINICAL TRIAL: NCT01031589
Title: Study in Healthy Volunteers to Examine the Safety, Tolerability and Plasma Pharmacokinetics of One Intramuscular (IM) Injection of a Novel TMC278 LA Formulation at 2 Different Doses (Open Label), Followed by a Placebo-controlled Part of Multiple IM Injections at a Selected Dose (Double Blind)
Brief Title: TMC278-TiDP15-C158 - A Study to Examine the Safety, Tolerability and Pharmacokinetics of a Single Dose or Three Successive Doses of Intramuscularly (IM) Injected Long Acting Formulation of TMC278
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR016747
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: HIV Infections
Keywords: TMC278-TiDP15-C158; TMC278-C158; TMC278; HIV; Non-nucleoside reverse transcriptase inhibitor; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Rilpivirine

INTERVENTIONS:
Drug: TMC278 (Rilpivirine) LA; Placebo

SUMMARY:
The purpose of this study is to examine the safety, local tolerability and pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) of a single intramuscular injection (injected directly in the muscle) of 300 mg (Panel 1) or 600 mg (Panel 2) of a new long acting form of TMC278. In Panel 3, the safety, local tolerability and pharmacokinetics are being studied after three successive intramuscular injections (single injection on Day1, single injection on Day15 and single injection on Day43) of a selected dose of the same TMC278 LA formulation. The dose of Panel 3 will be determined based on the safety, local tolerability and the pharmacokinetic results obtained in Panel 1 and 2.

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety, local tolerability and pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) of a newly selected long acting (LA) formulation of TMC278. This study will enroll 20 healthy volunteers. The first part of the study (Panel 1 + 2) is an open-label study (physician and volunteer know the identity of the drug that is injected) to determine the safety, tolerability and pharmacokinetics of a single IM injection of TMC278 LA. In the first Panel, 300 mg of TMC278 LA is injected once. After 3 days, if no safety or tolerability issues occur, a 600 mg dose of TMC278 LA is injected once in volunteers of Panel 2. The second part of the study is a double blind, placebo-controlled (neither physician nor the volunteer knows who is injected with TMC278 LA or placebo). Volunteers of this third Panel will receive 3 doses (one dose at Day 1, Day 15 and Day 43) of the same LA formulation of TMC278 as used in Panel 1 and 2. The Panel 3 dose will be selected based on the safety, tolerability and pharmacokinetic results obtained in Panel 1 and 2, which are being evaluated by a dedicated Data and Safety Review Committee. The dose for the three consecutive injections will be the same. In all Panels, the injections are given into the muscle of the buttock (alternating left and right buttock in Panel 3). Throughout the study, the injection sites will be monitored closely for signs of pain, pain at touch, itching, bruise, redness or other color, induration, swelling and inflammation by medical staff and the participating volunteers. Every Injection Site Reaction (ISR) that occurs will be documented as an adverse event. Additional safety assessments include monitoring of laboratory work including urine samples, vital signs and ECG. Volunteers of Panel 1 and 2 remain in follow-up for minimally 12 weeks after the injection. They are allowed to leave the study on condition that the TMC278 plasma concentration is below 20 ng/mL and that all previously emerged adverse events resolved or stabilized (i.e. according to the investigator and sponsor, the AE does not require further medical follow-up). The same conditions apply for volunteers of Panel 3. In Panel 1 and 2, volunteers receive one single IM dose of 300 mg or 600 mg TMC278 LA. In Panel 3, volunteers receive three IM doses consecutively (Day 1, Day 15 and Day 43) of TMC278 LA. The dose of the 3 injections in Panel 3 is to be determined, based on the safety, local tolerability and pharmacokinetic data of Panel 1 and 2. Six volunteers receive TMC278 LA, 2 receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker for at least 3 months prior to selection
* A BMI of 18.0 to 30.0 kg/m2
* Normal 12-lead electrocardiogram
* Healthy on the basis of physical examination, clinical laboratory tests, medical history and vital signs

Exclusion Criteria:

* Female, except if postmenopausal for at least 2 years or surgically sterile
* positive urine drug test
* History of clinically relevant skin disease or drug allergy
* Participation in an investigational drug study or having received a vaccine within 30 days prior to the first injection of TMC278 LA or placebo
* Previous participation in a study with oral TMC278, TMC125, TMC120 and/or TMC278 LA

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption of TMC278 following single or three successive IM injections | Panel 1 and 2 and after injection 2 and 3 in Panel 3: 672 hours; after injection 1 in panel 3: 336 hours.

SECONDARY OUTCOMES:
Results of Injection Site evaluations | Daily for the first week in the study, then weekly for minimally the next 12 weeks.
Safety Assessments (monitoring AEs, Lab, Vital Signs, ECG parameters) | Panel 1 and 2: Continuously throughout the 8 study visits; Panel 3: continuously throughout the 14 study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Derived] Verloes R, Deleu S, Niemeijer N, Crauwels H, Meyvisch P, Williams P. Safety, tolerability and pharmacokinetics of rilpivirine following administration of a long-acting formulation in healthy volunteers. HIV Med. 2015 Sep;16(8):477-84. doi: 10.1111/hiv.12247. Epub 2015 May 18. PMID 25988676